CLINICAL TRIAL: NCT04202783
Title: The Use of Exosomes In Craniofacial Neuralgia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending COVID-19 pandemic; pending product development
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICSS-2019-019
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: The present study is being undertaken as an open label study to evaluate the safety and feasibility of exosomes as an intervention for patients with craniofacial neuralgia. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures. The present study can be easily implemented because the neuropsychological testing instruments have been in routine clinical deployment providing for a high degree of availability and reliability. Quality assurance is tightly controlled. The study population is sufficiently broad and the conditions of interest are sufficiently prevalent so that recruitment of subjects is not a limiting factor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Craniofacial Neuralgia (Experimental): All patients will receive the same amount (5mL concentrated) of exosomes delivered via ultrasound-guided, regional epineural injection and the same amount (5mL unconcentrated) delivered via IV. Patients will be given 3 mL of the exosome product intravenously, which contains about 45mg of the exosome product containing 15-21 million neonatal stem cell products, and 3 mL of the exosome hyperconcentrate product delivered epineurally using ultrasound guidance, which contains about 15mg of the exosome product carrying 5-7 million neonatal stem cell products.
  Interventions: Other: Exosomes

INTERVENTIONS:
Other: Exosomes — Focused ultrasound delivery of intravenously-infused exosomes

SUMMARY:
This study is designed to evaluate the safety and efficacy of exosome deployment in patients with Craniofacial Neuralgia. Secondarily, this study is designed to rigorously evaluate for any adverse events that may be related to the administration and reception of exosomes.

DETAILED DESCRIPTION:
The present study is designed to amplify the delivery of growth factors and anti-inflammatory agents to localized targets (determined by specific condition) by using focused transcranial ultrasound prior to intravenous infusion of exosomes. Exosomes delivered intravenously can be demonstrated to cross the blood brain barrier naturally. Exosomes are thought to play a normal physiological role in intercellular signaling, and demonstrate anti-inflammatory and pro-growth effects in preclinical models and clinical cases reports. Clinical trials have deployed exosomes intravenously and with intracerebral and intrathecal injection, and have claimed safety and clinical efficacy.

Focused ultrasound has been shown to enhance local blood flow and has been presented as a non-invasive means of targeting delivery of therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Clinical diagnosis of craniofacial neuralgia

Exclusion Criteria:

* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Recent surgery or dental work within 3 months of the scheduled procedure.
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Any active cancer or chemotherapy
* Bone marrow disorder
* Myeloproliferative disorder
* Sickle cell disease
* Primary pulmonary hypertension
* Immunocompromising conditions and/or immunosuppressive therapies
* Macular degeneration
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced kidney, pulmonary, cardiac or liver failure
* Subjects with vascular causes of dementia
* Bleeding disorder, untreated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | 8 weeks from baseline
  The BPI is a 9 item self-report questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Patient Health Questionnaire (PHQ-9) | 8 weeks from baseline
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total possible score is 27 points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Adverse Event Reporting | Baseline to 24 weeks
  Adverse events (AEs) and any other untoward signs or symptoms were collected at each study timepoint starting at the treatment injection. Serious adverse events (SAEs) determined by the investigator to be related to the study treatment were formally recorded.

SECONDARY OUTCOMES:
Global Rating of Change (GRC) | 8 weeks from baseline
  The GRC is a self-administered one-item Likert scale questionnaire on the patient's overall satisfaction with the treatment; with scores from "-5" (very much worse) to "+5" (very much better). A GRC of at least is considered to be clinically significant improvement.
Brief Pain Inventory (BPI) | 24 weeks from baseline
  The BPI is a 9 item self-report questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Patient Health Questionnaire (PHQ-9) | 24 weeks from baseline
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total possible score is 27 points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Mikula I. [Craniofacial neuralgias]. Acta Med Croatica. 2008 May;62(2):163-72. Croatian. PMID 18710080
- [Background] Spina A, Mortini P, Alemanno F, Houdayer E, Iannaccone S. Trigeminal Neuralgia: Toward a Multimodal Approach. World Neurosurg. 2017 Jul;103:220-230. doi: 10.1016/j.wneu.2017.03.126. Epub 2017 Apr 2. PMID 28377244
- [Background] Rose FC. Trigeminal neuralgia. Arch Neurol. 1999 Sep;56(9):1163-4. doi: 10.1001/archneur.56.9.1163. No abstract available. PMID 10488822
- [Background] Cruccu G. Trigeminal Neuralgia. Continuum (Minneap Minn). 2017 Apr;23(2, Selected Topics in Outpatient Neurology):396-420. doi: 10.1212/CON.0000000000000451. PMID 28375911
- [Background] Maarbjerg S, Di Stefano G, Bendtsen L, Cruccu G. Trigeminal neuralgia - diagnosis and treatment. Cephalalgia. 2017 Jun;37(7):648-657. doi: 10.1177/0333102416687280. Epub 2017 Jan 11. PMID 28076964
- [Background] O'Neill F, Nurmikko T, Sommer C. Other facial neuralgias. Cephalalgia. 2017 Jun;37(7):658-669. doi: 10.1177/0333102417689995. Epub 2017 Jan 29. PMID 28133989
- [Background] Marchetti M, Pinzi V, De Martin E, Ghielmetti F, Fariselli L. Radiosurgery for trigeminal neuralgia: the state of art. Neurol Sci. 2019 May;40(Suppl 1):153-157. doi: 10.1007/s10072-019-03814-6. PMID 30838546
- [Background] Harding C, Heuser J, Stahl P. Receptor-mediated endocytosis of transferrin and recycling of the transferrin receptor in rat reticulocytes. J Cell Biol. 1983 Aug;97(2):329-39. doi: 10.1083/jcb.97.2.329. PMID 6309857
- [Background] Pan BT, Teng K, Wu C, Adam M, Johnstone RM. Electron microscopic evidence for externalization of the transferrin receptor in vesicular form in sheep reticulocytes. J Cell Biol. 1985 Sep;101(3):942-8. doi: 10.1083/jcb.101.3.942. PMID 2993317
- [Background] Johnstone RM, Adam M, Hammond JR, Orr L, Turbide C. Vesicle formation during reticulocyte maturation. Association of plasma membrane activities with released vesicles (exosomes). J Biol Chem. 1987 Jul 5;262(19):9412-20. PMID 3597417
- [Background] Bollini S, Gentili C, Tasso R, Cancedda R. The Regenerative Role of the Fetal and Adult Stem Cell Secretome. J Clin Med. 2013 Dec 17;2(4):302-27. doi: 10.3390/jcm2040302. PMID 26237150
- [Background] Balbi C, Piccoli M, Barile L, Papait A, Armirotti A, Principi E, Reverberi D, Pascucci L, Becherini P, Varesio L, Mogni M, Coviello D, Bandiera T, Pozzobon M, Cancedda R, Bollini S. First Characterization of Human Amniotic Fluid Stem Cell Extracellular Vesicles as a Powerful Paracrine Tool Endowed with Regenerative Potential. Stem Cells Transl Med. 2017 May;6(5):1340-1355. doi: 10.1002/sctm.16-0297. Epub 2017 Mar 8. PMID 28271621
- [Background] Zhang B, Yeo RW, Tan KH, Lim SK. Focus on Extracellular Vesicles: Therapeutic Potential of Stem Cell-Derived Extracellular Vesicles. Int J Mol Sci. 2016 Feb 6;17(2):174. doi: 10.3390/ijms17020174. PMID 26861305